CLINICAL TRIAL: NCT02588495
Title: Accuracy of Gastric Ultrasound to Diagnose a "Full Stomach". A Bayesian Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14-7883-BE
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Aspiration
Keywords: Ultrasound; Gastric area; Accuracy; Aspirate
MeSH Terms: interventions — Eating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasting (No Intervention): Participant will remain fasted following initial gastric ultrasound
- Food intake (Experimental): Participant will ingest either 250mL of clear fluid (apple juice) or 250mL of coffee and a muffin following initial gastric ultrasound
  Interventions: Other: Food intake

INTERVENTIONS:
Other: Food intake — Either drinking a cup of clear liquid, or having a cup of coffee and a muffin
  Arms: Food intake

SUMMARY:
During surgery, there is a risk that food or liquid in the stomach might be forced back up the throat where it could enter the lungs (aspirate) and result in serious complications or even death. This is why people going for surgery are required not to eat before their surgery. However, in emergency situations it is often not possible to know whether a patient has recently eaten or not. Anesthesiologists have recently developed an ultrasound test to determine if there is content in a patient's stomach and how much. This test involves an ultrasound examination of the abdomen and taking some measurements on the ultrasound screen.

The purpose of this study is to determine how accurate these measurements are. In other words, how good are we at detecting an empty stomach from one that has liquids, or solids in it. You are being asked to participate in this study because we require non-pregnant volunteers in order to answer the aforementioned study question.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 85 years
* Male or female
* American Society of Anesthesia physical status classification I and II
* Height greater than 145 cm
* Ability to understand the study protocol and provide informed consent

Exclusion Criteria:

* Subjects predisposed to have an increased residual gastric volume at baseline (eg. Diabetes or any known dysmotility)
* History of major upper gastrointestinal disease (including hiatus hernia or prior gastroduodenal surgery)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Ultrasound's sensitivity to identify a "full stomach" | 5 minutes
  Scanning the stomach to identify if the participant is fasted or has ingested liquid or solids

SECONDARY OUTCOMES:
Ultrasound's accuracy in detecting a "full stomach" | 5 minutes
  Assessing how accurate the Ultrasound machine is in detecting either liquid or solid contents in the participant's stomach after ingestion
Inter/Intra-rater reliability of observer in detecting a "full stomach" | 5 minutes
  Determining the reliability of observers in being able to similarly detect a full stomach

CONTACTS AND LOCATIONS:
Overall Officials: Anahi Perlas, MD, Principal Investigator — Staff Anesthesiologist
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530